CLINICAL TRIAL: NCT05148572
Title: Prospective Cohort Study of Changes in Circulatory MicroRNA After Surgical Resection of Hepatocellular Carcinoma (HCC) (PROSECT)
Brief Title: Prospective Cohort Study of Changes in Circulatory MicroRNA of Resected Hepatocellular Carcinoma
Acronym: PROSECT
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore Phenome Centre (Unknown); Nanyang Technological University (Other); MiRXES Pte Ltd (Industry); Asian Microbiome Library (AMiLi) Pte Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: AHCC11 PROSECT
Record Dates: First submitted 2021-11-16; First posted 2021-12-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma (HCC); Recurrence; miRNA biomarkers; Gut microbiota; Metabolites; Microbiome biomarkers; Circulating biomarkers
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples shall be used for relevant laboratory assessments. Blood, urine and stool samples shall be used for miRNA, microbiome and metabolome profiling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) is the 4th most common cause of cancer death globally but only 20% are diagnosed in its early stages where curative treatment can be carried out. Current standard-of-care surveillance of patients at high risk of developing HCC with 6-monthly serum alpha-fetoprotein (AFP) and ultrasound imaging (US) has a sensitivity of approximately 63% for detecting early HCC. There is an urgent need for a more efficacious and convenient modality of surveillance of high-risk patients to diagnose HCC at an early stage. In another study (AHCC10 ELEGANCE, NCT04965259), 2,000 patients at risk of developing HCC will be enrolled to develop the 1st miRNA in-vitro diagnostic (IVD) kit for HCC that has higher accuracy and better ease of use compared with the extant combination of AFP and US.

This prospective study will act as a positive control to the AHCC10 ELEGANCE Study and aims to address the absence of efficacious modalities of surveillance by validating a panel of circulating miRNA biomarkers signatures with histologically proven HCC. This study will determine progressive changes in the profiles of miRNA signatures pre- and post- surgical resection to identify signatures predictive of recurrence.

Additionally, this study also aims to identify changes in key metabolites and microbiome with correlation to changes in choline, bile acid and tryptophan metabolic pathways with changes in the composition and function of gut microbiota to establish actionable biomarkers that can predict HCC recurrence.

DETAILED DESCRIPTION:
This is a prospective study involving 100 patients with diagnosis of hepatocellular carcinoma (HCC) confirmed by histology at surgical resection. Eligible patients will receive CT scans at 6 months and 12 months post-surgery to monitor for recurrence. Pre- and post-surgery bio-samples (blood, urine, stool) will also be collected to monitor changes in profiles of miRNA, metabolome and microbiome.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female patients, 21 to 90 years of age at the time of signature of the informed consent form.
* The patient has clinically AND histologically proven HCC.
* The patient has R0 or R1 resection on histology.
* The patient has Child-Pugh <= 7 points without clinical ascites before surgery.
* The patient has ECOG performance status 0-1 before surgery.
* The patient is scheduled for liver resection within 6 weeks of signing screening informed consent form.
* The patient has received no anti-cancer specific treatment for HCC before the surgery (eg. previous liver resection, loco-regional therapy such as RFA, TACE, SIRT, radiotherapy, immunotherapy, chemotherapy or neo-adjuvant chemotherapy), other than the planned surgery. However, patient who has received previous HCC treatment more than 5 years ago is deemed to have a de-novo liver tumour and therefore can be included.
* The patient is able to comply with scheduled visits, assessments and other study procedures.
* The patient is willing to provide informed consent before enrolment in the study.

Exclusion Criteria:

* The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and highly likely to have been cured.
* The patient has active hepatic encephalopathy at time of enrolment.
* The patient has received a major organ allograft.
* The patient is known to be positive for the Human Immunodeficiency Virus (HIV).
* The patient has an uncontrolled bleeding disorder.
* The patient has uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or uncontrolled arrhythmia at the time of enrolment.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
* The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has received any investigational or non-registered medicinal product (drug or vaccine) within the 30 days preceding the date of enrolment.
* For female patients: the patient is pregnant or lactating.
* The patient is unable to provide informed consent or refuse blood taking.
* The patient has any other condition which, in the opinion of the Investigators, would make the patient unsuitable for enrolment or could interfere with completion of the study.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of hepatocellular carcinoma (HCC) confirmed by histology at surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
miRNA biomarker signatures diagnostic for HCC or for recurrence prediction. | Baseline and every 6 monthly thereafter, up to 12 months.
  Changes in the profile of circulating micro-RNA biomarkers pre- and post- surgical resection.
Gut microbiome profiling for recurrence prediction. | Baseline and every 6 monthly thereafter, up to 12 months.
  Differences in the profile of gut microbiota among HCC and healthy population retrieved from database.
Metabolome profiling for recurrence prediction. | Baseline and every 6 monthly thereafter, up to 12 months.
  Changes in the profile of metabolome in urine and plasma pre- and post- surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce CHOW, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (6):
- Singapore (6):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided